CLINICAL TRIAL: NCT01031316
Title: The Role of Serial Echocardiography to Detect an Asymptomatic Patent Ductus Arteriosus (PDA) in Very Low Birth Weight (VLBW) Infants: A Pilot Randomized Controlled Trial
Brief Title: Patent Ductus Arteriosus (PDA) Screening Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sara DeMauro, Assistant Professor of Pediatrics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 810241
Record Dates: First submitted 2009-12-01; First posted 2009-12-14 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Ductus Arteriosus, Patent
Keywords: Echocardiography; Infant, Premature; Infant, Very Low Birth Weight
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nondisclosure (Experimental)
  Interventions: Other: Nondisclosure of screening echocardiogram results
- Disclosure (Active Comparator)
  Interventions: Other: Disclosure of screening echocardiogram results

INTERVENTIONS:
Other: Nondisclosure of screening echocardiogram results — Subjects will be randomized to nondisclosure of screening echocardiogram results.
  Arms: Nondisclosure
Other: Disclosure of screening echocardiogram results — Subjects will be randomized to disclosure of screening echocardiogram results.
  Arms: Disclosure

SUMMARY:
The ductus arteriosus directs blood away from the pulmonary circulation and toward the systemic circulation during fetal life, then closes after birth. In preterm infants the incidence of spontaneous closure decreases with gestational age. Patent ductus arteriosus (PDA) increases the risks of bronchopulmonary dysplasia (BPD) and necrotizing enterocolitis (NEC). However, this association may not be a causal relationship.

Echocardiography is required to diagnose PDA. However, routine screening echocardiograms lead to detection of asymptomatic PDAs, for which the benefit of therapy remains unproven.

A randomized controlled trial has been designed in which 88 infants with birth weight less than or equal to 1250 grams and gestational age less than or equal to 30 weeks will be enrolled. The investigators' goal is to determine how screening echocardiography influences clinical management and outcomes in these infants.

ELIGIBILITY:
Inclusion Criteria:

* birth weight less than or equal to 1250 grams
* gestational age less than or equal to 30 weeks
* postnatal age less than or equal to 72 hours
* have a guardian or acceptable surrogate capable of giving consent on his/her behalf

Exclusion Criteria:

* not considered viable
* dysmorphic features or congenital malformations that adversely affect growth
* have known or suspected congenital heart disease (other than PDA)

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of days to regain birth weight. | 1-4 weeks

SECONDARY OUTCOMES:
Treatment for a PDA with indomethacin or surgical ligation. | 3-6 months
Necrotising enterocolitis (NEC) or >48 hours of NPO status for suspected NEC or feeding intolerance. | 3-6 months
Number of days to 120ml/kg/day of enteral feedings (full feeds). | 3-6 months
Ventilator days, number of days of positive airway pressure, and number of days in oxygen. | 3-6 months
Worst grade of intraventricular hemorrhage and presence of periventricular leukomalacia. | 3-6 months
Confirmed or suspected sepsis. | 3-6 months
Worst stage of retinopathy of prematurity. | 3-6 months
Day of death or discharge. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Schmidt, MD, Study Director — University of Pennsylvania/Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania